CLINICAL TRIAL: NCT04117100
Title: Advanced Endo-therapeutic Procedure : Registry-based Observational Study
Acronym: AE Registry
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Daniel Von Renteln, Gastroenterologist, Principal Scientist, MD, PhD, Centre hospitalier de l'Université de Montréal (CHUM)
Other Study IDs: 2018-7692/17.319
Record Dates: First submitted 2019-07-22; First posted 2019-10-07 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Zenker Diverticulum; Polyp of Colon; Colo-rectal Cancer
MeSH Terms: conditions — Zenker Diverticulum; Colonic Polyps; Colonic Neoplasms | interventions — Myotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Endoscopic mucosal resection (EMR): It has become the standard treatment for superficial tumors of the gastrointestinal tract, either flat or sessile: precancerous lesions and superficial cancers with no or low ganglionic risk. The pre-injection of physiological serum detaches the lesion from the deep plane and allows, with great security, the resection of the mucosa, muscularis mucosae with part of the submucosa, whatever the size and location of the lesion. Compared to other techniques, it allows a histological analysis which dictates the subsequent conduct and the possible need for a complementary surgery.
  Interventions: Procedure: Polypectomy or myotomy
- Endoscopic mucosal dissection (ESD): This technique uses submucosal injection and special knives to make a peri-lesional circumferential incision, followed by dissection through the submucosal sub-lesion.
  Interventions: Procedure: Polypectomy or myotomy
- Radio Frequency Ablation (RFA) and Argon Plasma Ablation (APC): This is a mucosal thermo-destruction technique. It uses a generator that delivers a sinusoidal current of high frequency to a probe covered with bipolar electrodes in tight network ensuring a uniform diffusion of the thermal effect. The tissue penetration is superficial on 1mm, intended to eradicate the epithelium up to the muscularis mucosae. Circumferential or focal probes are used as a function of the length of the segment to be treated.
  Interventions: Procedure: Polypectomy or myotomy
- Per Oral Endoscopic Myotomy (POEM): This technique allows a myotomy on the 8 cm of the lower esophagus extended on the gastric side of the cardia, totally endoscopically, after having approached and tunneled the esophageal submucosa.
  Less invasive, it gradually replaces the pneumatic dilatation and surgical myotomy of Heller.
  It requires a general anesthesia, an expert operator and a trained nursing team, ESD instruments, carbone dioxide insufflation.
  Interventions: Procedure: Polypectomy or myotomy

INTERVENTIONS:
Procedure: Polypectomy or myotomy — Advanced therapeutic endoscopy can replace surgery for treatment of benign and malign GI diseases and the aim of this registry-based study to improve quality related to advanced therapeutic endoscopy because the trial will provides a quantitative method to assess advanced therapeutic practise at the CHUM and may identify practices of low quality (possible intervention) or high quality (desired). Advanced therapeutic endoscopy procedures included for this registry-based study are EMR, ESD, Assessment of polypectomy quality for colorectal adenomas/polyps, Radio Frequency Ablation (RFA) and Argon Plasma Ablation (APC), and Per Oral endoscopic Myotomy (POEM).

SUMMARY:
Advanced therapeutic endoscopy procedures are of increasing importance to provide minimal invasive treatment for GI diseases. The Centre Hospitalier de l'Université de Montréal as tertiary university center is dedicated to increase the availability of therapeutic endoscopy procedures for our population in Montreal and Quebec. Advanced endotherapeutic endoscopy can replace surgery for treatment of benign and malign GI diseases and the aim of this registry-based study is to improve quality related to advanced endotherapeutic endoscopy, as it will provide quantitative means to assess advanced endotherapeutic practice and may identify practices of low quality (possible intervention) or high quality (desired).

DETAILED DESCRIPTION:
Advanced therapeutic endoscopy procedures included for this registry-based study are endoscopic mucosal resection (EMR), Endoscopic mucosal dissection (ESD), Assessment of Polypectomy quality for colorectal adenomas/polyps, Radio frequency Ablation (RFA) and Argon Plasma Ablation (APC), and Per Oral endoscopic Myotomy (POEM). All patients who present for an advanced endotherapeutic endoscopy (ESD, EMR, deep resection, POEM or Zenker treatment) may be included into the registry. Data will be collected prospectively. Data will be recorded on case report forms (CRF), which will then be transferred to an electronic data base (= registry), located on a protected drive.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Presenting for an elective advanced therapeutic endoscopy (ESD, EMR, advanced polypectomy, POEM or Zenker treatment)
* Signed informed consent form

Exclusion Criteria:

* Patients that are not capable understanding the trial and patients without consent.
* Patients with coagulopathy
* Patient with poor general health defined as an American Society of Anesthesiologists class greater than three
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible participants presenting at the CHUM for an elective advanced therapeutic endoscopy (ESD, EMR, advanced polypectomy, POEM or Zenker treatment) will be approached for this research project.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence of overall severe complications following the procedure | 14 days
  Aggregate of all severe adverse events that occur at the time of the procedure (immediate complications) or during 14 days of follow-up. Severe adverse events include bleeding, perforation, and clinical events that require an admission to the hospital.
Assess the rate of completeness of neoplastic tissue resection | 6-18 months
  Assessment of the complete adenoma/Barretts/dysplastic tissue removal, defined as removal of all visible neoplastic tissue at the end of the EMR as assessed by the endoscopist.
Severe bleeding complications | 14 days
  Immediate or delayed: severe bleeding is defined as the need for hospitalization, transfusion, a repeat endoscopy, surgery, or interventional radiology. An immediate complication is defined as an event at the time of resection or immediately following the endoscopy (before patient has left the endoscopy unit/during immediate post-colonoscopy care). A delayed complication is defined as a bleeding event that occurred after the patient has left the endoscopy unit and within 14 days following the procedure.
Assess the presence of perforation at resection site | 6-18 months
  Assessment of the presence of a complete hole, or full-thickness resection of the muscularis propria
Assess the number of patients with post-polypectomy syndrome | 6-18 months
  As defined as abdominal pain severe enough to warrant an ER visit or hospital admission and presence of leukocytosis and/or required treatment with antibiotics.
Assess the efficacy of submucosal injectate | 6-18 months
  Assessment of the solution volume per lesion size (ml/cm2), time of resection.
Assess the number of patients with intraprocedural bleeding | 6-18 months
  Assessment of immediate bleeding that requires endoscopic intervention to stop the bleeding (e.g. clip placement or snare tip soft coagulation or coagulation grasper).
Assess the number of patients with the need for surgical resection | 6-18 months
  Assessment of patients that require surgery for removal of precancerous or cancerous lesions or as result of complications related to the EMR/ESD or endoscopy intervention or for follow-up procedures.
Technical skill of the endoscopist | 6-18 months
  Video based assessment of endoscopic resection skills
En-bloc resection rate | 6-18 months
  The number of cases with complete removal of the targeted lesion in a single piece without fragmentation (ensuring the entire specimen can be assessed for histopathological margins and integrity) out of all the cases.
R0 resection rate | 6-18 months
  The number of cases with a resection with histologically confirmed negative margins (indicating no residual tumor cells at the resection site, both lateral and deep margins are free of neoplastic involvement) out of all cases.
Local recurrence rate | 6-18 months
  The rate of reappearance of biopsy-confirmed neoplastic tissue at the original resection site during surveillance endoscopies or detection of cancer in the same area on imaging after the initial curative treatment.
Distant metastasis rate | 6-18 months
  The rate of development of cancerous spread to distant organs or sites beyond the original tumor location after initial curative treatment.
Lymph node involvement rate | 6-18 months
  The rate of detection of cancerous infiltration in regional or distant lymph nodes, identified through imaging, biopsy, or surgical pathology, after initial curative treatment.
Disease progression | 6-18 months
  Worsening of the disease, as evidenced by local recurrence, distant metastasis, lymph node involvement, or the appearance of new lesions, after the initial curative treatment.
Progression-free survival (PFS) | 6-18 months
  The time from the date of initial treatment to the earliest occurrence of disease progression (local recurrence, distant metastasis, lymph node involvement, or new lesion development) or death from any cause, whichever occurs first.
Cancer-related mortality | 6-18 months
  Death directly attributable to the primary cancer or its complications, as determined by clinical assessment, autopsy, or death records.
All-cause mortality | 6-18 months
  Death from any cause, including cancer-related and unrelated causes, during the study period or follow-up after initial curative treatment.
Time to recurrence | 6-18 months
  The interval between the date of initial curative treatment and the detection of local recurrence or distant metastasis.
Quality of life (QoL) score | 6-18 months
  Patient-reported or clinician-assessed outcomes measuring physical, emotional, and social well-being, as well as symptom burden, during or after treatment. The EQ-5D-5L score will be used, which is a health status measurement that ranges from -0.59 to 1, where 1 indicates excellent health status.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, MD,PhD, Principal Investigator — Centre Hospitalier Universitaire de Montréal (CHUM)
Locations (1):
- Centre Hospitalier Universitaire de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided